CLINICAL TRIAL: NCT02278549
Title: Comparison of Spinal Kinematics Between Asymptomatic Subjects and Patients With Low Back Pain Using a Multi-segment Model
Brief Title: Comparison of Spinal Kinematics Between Asymptomatic Subjects and Patients With Low Back Pain
Status: Completed | Type: Observational
Sponsor: Haute Ecole de Santé Vaud (Other)
Collaborators: University of Brighton (Other); University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Guillaume Christe, PT, Haute Ecole de Santé Vaud
Other Study IDs: MT001GC
Record Dates: First submitted 2014-10-27; First posted 2014-10-30 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Low Back Pain
Keywords: Spinal kinematics
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Asymptomatic: Individuals between 30 and 50 years old that have had no episode of low back pain in the last two years requiring medical attention
- Patients with Low Back Pain: Individuals between 30 and 50 years old that present with non-specific low back pain for more than 3 months

SUMMARY:
Low back pain (LBP) is a complex and common problem with major societal repercussions. Clinical evaluations, and especially functional assessments, are necessary for proper diagnosis and decisions on the most appropriate treatment. The assessment of lumbar kinematics has been frequently described. For instance, measures of range of motion (ROM), angular velocities and acceleration of the total lumbar spine (TLx) have demonstrated some differences between healthy subjects and LBP patients. However, recent evidence has suggested that models evaluating the TLx are insufficient. In fact, regional differences in kinematics have been described between the upper lumbar spine and the lower lumbar spine.

The aim of this study is to evaluate the differences in spinal kinematics between healthy subjects and LBP patients using a multi-segment model of the spine that allows regional analysis.

DETAILED DESCRIPTION:
A case-controlled study will be performed to compare asymptomatics subjects and patients with low back pain. ROM, angular velocities and coordination of the spine will be collected in a laboratory with a camera-based system (VICON). Subjects will have to perform normal ROM assessment in the three anatomical planes, as well as different functional activities such as sit to stand, step and walking. The measurement session will occur on one occasion for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient French level
* BMI between 18 and 27
* Non-specific low back pain for more than 3 months (pain provoked by movements, postures or activities)

Exclusion Criteria:

* Pregnancy
* Spondylolisthesis
* Infection
* Rheumatological or neurological diseases
* Spinal fractures
* Known spinal deformation (scoliosis, …)
* Back surgery
* Tumours
* Radicular symptoms (with neurological signs). Pain irradiating in the lower limbs with decrease strength, sensitivity and reflex.
* High level of pain (severity and irritability) at the time of experiment that prevents repeated movements.
* Other concomitant pain or condition that could compromise the evaluation of lumbar kinematics.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with recurrent low back pain (more than months in duration) recruited through physiotherapy practices and medical consultations in the area of Lausanne, Switzerland.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Spinal kinematics | Participants will be measured once
  kinematics of the spine and pelvis will be measured with a camera-based system. Markers will be placed to have different segments of the spine (lower lumbar spine, upper lumbar spine, lower thoracic spine, upper thoracic spine). Variables such as range of motion, angular velocities or coordination (among others) will be measured.

SECONDARY OUTCOMES:
Score of disability | Participants will be measured once
  Oswestry Disability Index. Outcome used primarily for description of the population and correlational analysis
Score of kinesophobia | Participants will be measured once
  Tampa Scale of kinesophobia. Outcome used primarily for description of the population and correlational analysis
Score of risk of poor outcomes | Participants will be measured once
  Start Back Tool. Outcome used primarily for description of the population and correlational analysis
Pain intensity | Participants will be measured once
  Numeric Pain Rating Scale (NPRS). Outcome used primarily for description of the population and correlational analysis

CONTACTS AND LOCATIONS:
Overall Officials: Julien Favre, PhD, Study Director — University of Lausanne Hospitals; Lucy Redhead, PhD, Study Director — University of Brighton; Guillaume Christe, PT, Principal Investigator — Haute Ecole de Santé Vaud
Locations (1):
- University of Lausanne Hospitals, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Cobian DG, Daehn NS, Anderson PA, Heiderscheit BC. Active cervical and lumbar range of motion during performance of activities of daily living in healthy young adults. Spine (Phila Pa 1976). 2013 Sep 15;38(20):1754-63. doi: 10.1097/BRS.0b013e3182a2119c. PMID 23823575
- [Background] Crosbie J, Nascimento DP, Filho Rde F, Ferreira P. Do people with recurrent back pain constrain spinal motion during seated horizontal and downward reaching? Clin Biomech (Bristol). 2013 Oct;28(8):866-72. doi: 10.1016/j.clinbiomech.2013.09.001. Epub 2013 Sep 9. PMID 24067874
- [Background] Dankaerts W, O'Sullivan P, Burnett A, Straker L. Differences in sitting postures are associated with nonspecific chronic low back pain disorders when patients are subclassified. Spine (Phila Pa 1976). 2006 Mar 15;31(6):698-704. doi: 10.1097/01.brs.0000202532.76925.d2. PMID 16540876
- [Background] Lehman GJ. Biomechanical assessments of lumbar spinal function. How low back pain sufferers differ from normals. Implications for outcome measures research. Part I: kinematic assessments of lumbar function. J Manipulative Physiol Ther. 2004 Jan;27(1):57-62. doi: 10.1016/j.jmpt.2003.11.007. PMID 14739876
- [Background] Marras WS, Ferguson SA, Gupta P, Bose S, Parnianpour M, Kim JY, Crowell RR. The quantification of low back disorder using motion measures. Methodology and validation. Spine (Phila Pa 1976). 1999 Oct 15;24(20):2091-100. doi: 10.1097/00007632-199910150-00005. PMID 10543004
- [Background] Parkinson S, Campbell A, Dankaerts W, Burnett A, O'Sullivan P. Upper and lower lumbar segments move differently during sit-to-stand. Man Ther. 2013 Oct;18(5):390-4. doi: 10.1016/j.math.2013.02.001. Epub 2013 Mar 7. PMID 23473753
- [Background] Wade M, Campbell A, Smith A, Norcott J, O'Sullivan P. Investigation of spinal posture signatures and ground reaction forces during landing in elite female gymnasts. J Appl Biomech. 2012 Dec;28(6):677-86. doi: 10.1123/jab.28.6.677. Epub 2012 May 10. PMID 22661081